CLINICAL TRIAL: NCT06016517
Title: Application of the Personalized N-of-1 Trial Design in Patients With Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00003917
Record Dates: First submitted 2023-06-26; First posted 2023-08-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab; upadacitinib; tocilizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Etanercept — 50 mg subcutaneously weekly
  Other Names: Enbrel
Drug: Adalimumab — 40 mg subcutaneously every 2 weeks
  Other Names: Humira
Drug: Upadacitinib — 15 mg orally once daily with subcutaneous placebo injection every 2 weeks
  Other Names: Rinvoq
Drug: Tocilizumab — 162 mg administered SQ every 2 weeks

SUMMARY:
The goal of this N-of-1 study is to learn about treatment for individual patients who have rheumatoid arthritis (RA,) for which many treatments are available. The treatments are different in how they work, the way they are given, side- effects, and cost. While treatment guidelines are available, finding the best treatment order of treatments is often based on physician choice. The main question this study aims to answer are:

* What are the effects of different treatments on RA symptoms and condition for each individual patient
* What is the effectiveness of different treatments across all patients enrolled in the N-of-1 study

Participants will be enrolled and randomized to a sequence of three U.S. Food and Drug Administration (FDA) approved RA medications: 1. etanercept, 2. adalimumab, 3. upadacitinib 4. tocilizumab. Participants will be asked to complete questionnaires about their condition and quality of life fortnightly, monthly and/or quarterly (either in clinic or remotely) and report their level of pain on alternate days (remotely).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, slowly progressive condition for which numerous treatment options are available. The therapies vary in mechanism of action, mode of administration, side- effect (adverse event) profile, and cost. While consensus treatment guidelines are available, identifying an optimal treatment sequence is often based on clinician choice with treatment changes based on tolerability and short- term outcome. The N-of-1 trial will evaluate individual participant and aggregate data.

Individual participants will be enrolled and randomized to a sequence of three U.S. Food and Drug Administration (FDA)-approved therapeutic agents etanercept, adalimumab, upadacitinib and tocilizumab.

The N-of-1- RA protocol describes patient allocation into a series of individual comparisons.

• Patients with newly diagnosed rheumatoid arthritis following initial treatment with methotrexate (MTX). Participants will be allocated to:

* MTX responder
* MTX non- responder or partial responder

Eligible participants will either continue MTX or discontinue MTX, based on response to initial therapy and tolerance. Participants identified for subsequent biologic therapy will enter the biologic therapy phase of the study; with MTX either continued or not continued. This phase consists of a sequence of 4 therapeutic intervention regimens, each lasting 12-weeks.

The treatment conditions are as follows:

A. Tumor Necrosis Factor (TNF) Inhibitor biologic: etanercept 50 mg subcutaneously weekly.

B: TNF- inhibitor biologic: Adalimumab 40 mg subcutaneously every 2 weeks. C. Janus Kinase (JAK) Inhibitor: Upadacitinib 15 mg orally once daily. D. Interleukin 6 (IL-6) Inhibitor: Tocilizumab 162 mg administered SQ every 2 weeks (if there is an inadequate response to prior three biologics).

Primary Objective (individual N-of-1 trial): To generate randomized evidence about the effects of therapeutic agents on RA symptoms and disease activity to inform decision about best treatment at the end of the trial period for each participant.

Secondary Objective (aggregation of the series of N-of-1 trials): To evaluate the average relative effectiveness of therapeutic agents across all participants and explore heterogeneity of treatment effects.

For the aggregated series of N-of-1 trial, we will use the following hierarchy of endpoints.

Primary Endpoint:

• DAS28 (CRP and ESR)

Secondary Endpoints:

* American College of Rheumatology 20% (ACR20), 50% (ACR50) and 70% (ACR70) response
* Routine Assessment of Patient Index Data (RAPID3) score based on participants' report of overall assessment of the disease, the level of pain, and the amount of physical disability
* Short Form 12-Item Health Survey (SF-12) measuring the impact of disease on overall quality of life during the prior 4 weeks (physical function, pain, general and mental health, vitality, social function, physical and emotional health)
* Report of worst pain and effect of pain on function (0-10) every other day
* Treatment Burden Questionnaire (TBQ) administered at the end of each treatment condition

Safety Endpoint(s):

• Number (and proportion) of patients reporting treatment emergent adverse events (TEAEs) (by MedDRA system organ class and preferred term)

For each individual N-of-1 trial, we will use the endpoints listed above, but without any pre-specified hierarchy, assuming that each patient will identify endpoints most important to them.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all the following criteria:

* Newly diagnosed adult-onset Rheumatoid Arthritis (RA) as defined by the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2021 Criteria for the Classification of RA
* Moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* C-reactive protein (CRP) or high-sensitivity C-reactive protein (hsCRP) measurement ≥ 1 time the upper limit of normal
* First-line therapy with MTX for at least the 12 weeks prior to study entry with a continuous, non-changing dose for at least 8 weeks prior to study entry but continue to exhibit active RA
* Had to discontinue MTX due to intolerability or toxicity, irrespective of treatment duration
* Have never received etanercept, adalimumab, upadacitinib, or tocilizumab prior to first dose of study drug.
* Provision of informed consent in English or another language in which a validated consent form is available, or via short-form consent with the assistance of a qualified interpreter.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 18 years of age or older
* Ability to take oral medication and be willing to adhere to all treatment periods
* Patients are eligible whether their disease responded partially or inadequately to first-line MTX or if they were intolerant to first-line MTX
* Enrollment in an insurance plan that participates in or is subscribed to this trial

An individual who meets any of the following criteria will be excluded from participation in this study:

* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA
* Has received intra-articular, intravenous, intramuscular corticosteroids within 28 days prior to baseline
* Known allergic reactions to components of any of the investigative biologic agents
* Is currently receiving corticosteroids at doses > (greater than) 10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization
* Has experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or have New York Heart Association stage IV heart failure
* Tuberculosis infection
* Hepatitis B or C infection
* History of venous thromboembolic event (deep vein thrombosis, pulmonary embolism)
* Has a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk or could interfere with the interpretation of data
* Has an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine of < (less than) 40 milliliter per minute per 1.73 m^2 (mL/min/1.73 m^2)
* Has a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin ≥1.5 times the ULN
* Has a history of, lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years
* Has been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination)
* Has a current or recent clinically serious viral, bacterial, fungal, or parasitic infection
* Has had symptomatic herpes zoster infection within 12 weeks prior to study entry
* Has immunocompromising condition and, in the opinion of the investigator, are at an unacceptable risk for participating in the study and using these medications
* Has a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)*
* Has evidence of active or latent tuberculosis (TB)
* Current hospitalization or requiring hospital admission at screening
* Pregnant or breastfeeding
* Of childbearing potential, unwilling to use effective birth control method (highly effective contraceptive measure (e.g., combined (estrogen and progestogen containing) hormonal contraception; intrauterine device)
* Participation in another therapeutic clinical trial for RA
* Lack of internet access to telehealth platform

State who will determine eligibility. Note that those who are designated to determine eligibility must have appropriate training, expertise, and oversight, for example a physician PI or Co-I on a biomedical study: Eligibility will be determined by the appropriately trained and delegated physician investigator or physician Co- investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients 18 years of age or older with newly diagnosed RA following initial treatment with MTX, to which they are partial responders or non-responders.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Disease Activity Score (DAS) 28 | Baseline and week 12 of each treatment period
  Evaluates patient and physician overall assessment of disease activity, including the number of swollen and painful joints (out of 28 joints),

SECONDARY OUTCOMES:
Change in The Routine Assessment of Patient Index Data 3 (RAPID3) | Baseline, and weeks 2, 4, 6, 8, 10, 12 of each treatment period
  Assessment of a) function, b) pain, and c) patient global estimate of status
Change in American College of Rheumatology 20 (ACR20) | Baseline and week 12 of each treatment period
  ≥20% fewer tender and swollen joints and ≥20% improvement in three of five other domains; a) patient global assessment, b) physician global assessment, c) functional questionnaire, d) pain score, and f) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)
Change in American College of Rheumatology 50 (ACR50) | Baseline and at week 12 of each treatment period
  ≥50% fewer tender and swollen joints and ≥20% improvement in three of five other domains; a) patient global assessment, b) physician global assessment, c) functional questionnaire, d) pain score, and f) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)
Change in American College of Rheumatology 70 (ACR70) | Baseline and at week 12 of each treatment period
  ≥70% fewer tender and swollen joints and ≥20% improvement in three of five other domains; a) patient global assessment, b) physician global assessment, c) functional questionnaire, d) pain score, and f) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)
The Medical Outcome Study Short-Form 12- item Health Survey (SF-12) | Baseline and at week 4, 8, and 12 of each treatment period
  General Health Questionnaire
Treatment Burden Questionnaire (TBQ) | At week 36
  Assessment of the burden associated with taking medicine, self-monitoring, laboratory tests, doctor visits, need for organization, administrative tasks, following advice on diet and physical activity, and social impact of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Harry P Selker, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States